CLINICAL TRIAL: NCT03963674
Title: Effects of Diacutaneous Fibrolysis Over the Gastrocnemious Neuromuscular Response
Brief Title: Effects of Diacutaneous Fibrolysis Over Neuromuscular Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Principal investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol 5
Record Dates: First submitted 2019-05-20; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-02

CONDITIONS: Myofascial Pain Syndrome; Contraction
Keywords: Neuromuscular response; diacutaneous fibrolysis
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diacutaneous fibrolysis (Experimental)
  Interventions: Other: Diacutaneous fibrolysis
- Control (No Intervention)

INTERVENTIONS:
Other: Diacutaneous fibrolysis — Diacutaneous fibrolysis over the gastrocnemious muscles
  Arms: Diacutaneous fibrolysis

SUMMARY:
The study consists in evaluating the neuromuscular response of the gastrocnemious muscles before and after a diacutaneous fibrolysis over the gastrocnemious muscles.

ELIGIBILITY:
Exclusion Criteria:

* Muscle injury in the last two months
* To not understand the study orders
* Suffer a musculoskeletal disorder that doesn't allow the subject to do the study protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-06-05 (Estimated)

PRIMARY OUTCOMES:
Delay time change | 4 minutes before the intervention, 5 minutes after the intervention and 30 minutes later
  Time between an electric impulse and 10% of the contraction of the muscle that is being excited with an electric impulse, using an electromyography test (miliseconds).
Contraction time change | 4 minutes before the intervention, 5 minutes after the intervention and 30 minutes later
  Time between 10% and 90% of the contraction of the muscle that is being excited with an electric impulse, using an electromyography test (miliseconds).
Sustain time change | 4 minutes before the intervention, 5 minutes after the intervention and 30 minutes later
  time between 50% of the contraction and 50% of the relaxation of the muscle after being impulsed with an electric impulse, using an electromyography test (miliseconds).
Relaxation time change | 4 minutes before the intervention, 5 minutes after the intervention and 30 minutes later
  time between 90% and 50% of the relaxation of the muscle after being impulsed with an electric impulse, using an electromyography test (miliseconds).
Maximal displacement change | 4 minutes before the intervention, 5 minutes after the intervention and 30 minutes later
  Maximal displacement of the muscle after being excited with an electric impulse, using an electromyography test (miliseconds).
Stiffness change | 2 minutes before the intervention, 7 minutes after the intervention and 30 minutes later
  Resistance to an external force that deforms its initial shape, using a "Myoton" (Newtons/metre).
Elasticity change | 2 minutes before the intervention, 7 minutes after the intervention and 30 minutes later
  Capacity to recover its initial shape after the removal of the external force that lead to its deformation, using a "Myoton" (logarithmic decrement of a tissue's natural oscillation).
Relaxation change | 2 minutes before the intervention, 7 minutes after the intervention and 30 minutes later
  Time for a muscle to recover its shape from deformation after the removal of an external force, using a "Myoton" (miliseconds).

SECONDARY OUTCOMES:
Gastrocnemious strength change | 8 minutes before the intervention, 1 minute after the intervention and 30 minutes later
  Isometric strength of the gastrocnemious muscles using a handheld dynamometer "microFET 2" (newtons).

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Pérez-Bellmunt, Sant Cugat del Vallès, Barcelona, Spain